CLINICAL TRIAL: NCT05973903
Title: Lenvatinib, Pembrolizumab, and Tumor Treating Fields (TTFields) for Second-line Treatment of Glioblastoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: It was decided by the researcher not to open the study due to administrative issues.
Sponsor: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, Deborah T. Blumenthal, MD, Director of Neuro-Oncology Tel-Aviv Sourasky Medical Center, Tel Aviv Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0489-22 TLV
Record Dates: First submitted 2023-07-20; First posted 2023-08-03 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: GBM
MeSH Terms: interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Forty-seven patients will be included in the study: 10 patients as "lead-in" (phase I) and 37 patients in phase II.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Single-arm: participants will be treated with TTFields (200 kHz) + intravenous pembrolizumab 200 mg every three weeks and oral lenvatinib 20 mg once daily until evident progressive disease by Response Assessment in Neuro-Oncology (RANO) criteria, unacceptable toxicity, withdrawal of consent, or until completion of 35 treatment cycles (approximately 2 years) with pembrolizumab. Participants who complete treatment with pembrolizumab after 35 cycles (approximately 2 years) or CR will continue to receive lenvatinib and TTF until disease progression, development of unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab; Device: Tumor Treating Fields (TTFields)

INTERVENTIONS:
Drug: Lenvatinib — Oral Lenvatinib 20 mg once daily
  Other Names: LENVIMA®, KISPLYX®
Drug: Pembrolizumab — intravenous pembrolizumab 200 mg every three weeks
  Other Names: Keytruda
Device: Tumor Treating Fields (TTFields) — TTF extra-dermal scalp electrodes

SUMMARY:
This will be a prospective, open label, single center, phase I lead-in study of 10 patients to a single arm phase-II study of 37 additional patients to assess the effectiveness of pembrolizumab and lenvatinib combination therapy for recurrent glioblastoma (rGBM) patients wearing TTFields electrodes.

DETAILED DESCRIPTION:
Male and female patients, 18 years of age or older, with confirmed GBM progressed after first-line treatment. Patients either with or without first-line TTFields alternating field therapy - will be eligible to enroll in the study.

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or legally acceptable representative if applicable) provided written informed consent for the trial.
2. Males and females at least 18 years of age on the day of signing informed consent with histopathologic evidence of GBM (from original or recurrent diagnosis) and MRI-confirmed diagnosis of rGBM.
3. Have received front-line treatment (chemo-radiation with temozolomide with or without adjuvant monthly temozolomide, with or without TTF with first line therapy) per local standard of care or treatment guideline following the primary surgery with radiologically documented disease recurrence after first-line therapy.
4. Wears TTFields electrodes or is suitable for wearing TTFields electrodes.
5. A predicted life expectancy of >3 months.
6. Have Karnofsky Performance Status (KPS) ≥70% (ECOG 0-1).
7. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 120 days (corresponding to the time needed to eliminate any study treatments) after the last dose of study treatment and refrain from donating sperm during this period.
8. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days (corresponding to time needed to eliminate any study treatments) after the last dose of study treatment.
9. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of the tumor lesion.

   Note: Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.

   Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
10. Have adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg at Screening and no change in antihypertensive medications within 1 week before the first dose of study treatment.
11. Have adequate organ function as defined in Table 1 below. Specimens must be collected within 10 days prior to the start of study treatment

Exclusion Criteria:

1. Has an implanted pacemaker, defibrillator, deep brain stimulator, other implanted electronic devices in the brain.
2. Has evidence of increased intracranial pressure (midline shift >5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness).
3. A WOCBP who has a positive urine pregnancy test within 72 hours prior to enrollment (see Appendix 3) as documented by a positive beta-human chorionic gonadotropin [Beta-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 IU/L or equivalent units of Beta-hCG [or hCG]). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
4. Is pregnant or breastfeeding at Screening or Baseline or expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
5. Has received prior therapy with an anti-PD-1, anti-PD-L1 or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) in the last 6 months (6 months are calculated from the last dose until study initiation).
6. Has received prior systemic anti-cancer therapy mAb, chemotherapy or targeted small molecule therapy within 4 weeks prior to the planned first dose of the study, including investigational agents within 4 weeks. For tyrosine kinase inhibitors (TKIs) and hormonal therapy a shorter interval of 5 half-lives is allowed between prior therapy and study treatment initiation.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: If the participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment. Do not administer lenvatinib for at least 2 weeks following major surgery and until adequate wound healing.
7. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, and not have had radiation pneumonitis.
8. Had prior grade 3 immune-related toxicity due to immune checkpoint inhibitors or non-infectious pneumonitis.
9. Has a history of active tumor bleeding one month before study enrollment.
10. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Note: mRNA vaccination for SARS-CoV-2 is not an exclusion.
11. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. (Note: subjects who participated in local TTF study #0412-08 [A prospective, multi-center trial of NovoTTF-100A together with temozolomide (TMZ) compared to TMZ alone in patients with newly diagnosed glioblastoma (GBM)] and are in follow-up may be eligible for the current study). Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
12. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 2 mg daily dexamethasone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

    Note: The use of physiologic doses of corticosteroids is allowed.
13. Has a known active second/additional malignancy that is progressing or has required active treatment within the past 5 years Note: Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy.
14. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or lenvatinib and/or any of their excipients.
15. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

    Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
16. Has an active infection requiring systemic therapy.
17. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
18. Has a known history of human immunodeficiency virus (HIV 1/2 antibodies).
19. Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as detected qualitative HCV RNA) infection.

    Note: no testing for hepatitis B and hepatitis C is required unless a known history of infectious hepatitis is reported.
20. The participant has a known history of active Bacillus Tuberculosis (TB).
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
22. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. Has had an active allogenic tissue/solid organ transplant.
24. Has uncontrolled blood pressure (Systolic BP>150 mmHg or diastolic BP>90 mmHg) despite an optimized regimen of antihypertensive medication during 7 days prior to starting study treatment, or the participant has adequately-controlled blood pressure but has had a change in antihypertensive medications within 7 days before the first dose of study treatment.
25. Has clinically significant electrolyte abnormalities that have not been corrected.
26. Has significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction (MI) or cerebrovascular accident (CVA) within 6 months of the first dose of study drug, or cardiac arrhythmia associated with hemodynamic instability requiring medical treatment at Screening.
27. Has bleeding or thrombotic disorders, radiographic evidence of major blood vessel invasion/infiltration, or is at risk for severe hemorrhage.

    Note: The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
28. Has >1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
29. Has prolongation of QTc interval to >480 ms.
30. Has left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO).
31. Has gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
32. Has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula.
33. Has a known intolerance to the study treatment (or any of its excipients).

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS-6) | 6 months
  Treatment with pembrolizumab and lenvatinib in rGBM patients wearing TTFields electrodes is expected to increase PFS-6 from 15 to 30%.

IPD SHARING:
Plan to Share IPD: No